CLINICAL TRIAL: NCT01897181
Title: Evaluation of the Central Auditory Processing in Patients (Elder Than 45 Years Old) With Bilateral Sensorineural Hearing Loss and the Change of the Central Auditory Processing Ability by the Use of Hearing Aids (CAPHA)
Brief Title: Central Auditory Processing and the Use of Hearing Aids
Acronym: CAPHA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jong Woo Chung (Other)
Responsible Party: Sponsor-Investigator, Jong Woo Chung, MD, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AMC-2013-0455
Record Dates: First submitted 2013-07-05; First posted 2013-07-11 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Auditory Processing Disorder, Central
Keywords: Central auditory processing; Bilateral sensorineural hearing loss; Hearing aids
MeSH Terms: conditions — Language Development Disorders | interventions — Hearing Aids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hearing aids (Active Comparator): Patients who agree to use hearing aids
  Interventions: Device: Hearing aids
- No hearing aids (No Intervention): Patients who did not agree to use hearing aids

INTERVENTIONS:
Device: Hearing aids — Using hearing aids for 12 months
  Arms: Hearing aids

SUMMARY:
The purpose of this study is to evaluate the central auditory processing in patients with bilateral sensorineural hearing loss and to observe the change of the central auditory processing ability after using hearing aids.

DETAILED DESCRIPTION:
Screening for recruiting

* Among patients who are visiting for hearing disturbance, patients with bilateral sensorineural hearing loss will be included after audiologic tests, history taking and physical examination.
* audiologic tests: pure tone audiometry, speech audiometry, impedence audiometry, distortion product otoacoustic emission, auditory brainstem response.

Dividing into "Hearing aids" group and "No hearing aids" group

* The use of hearing aids will be recommended to all included patients.
* Hearing aids group: patients who want to be prescribed hearing aids (28 subjects)
* No hearing aids group: patients who do not want to be prescribed hearing aids (28 subjects)

Audiologic test

* Hearing in noise test (HINT), central auditory processing disorder test
* at screening, 1, 3, 6, 9 and 12 months after starting hearing aids use

ELIGIBILITY:
Inclusion Criteria:

* Adults of age 45 years of older
* Bilateral sensorineural hearing loss
* Average pure tone audiometry threshold >= 40dB
* Speech discrimination >= 60% in both ears

Exclusion Criteria:

* Refusing the study
* Medical history of any brain damage or intracranial surgery
* Showing signs of central lesion in MRI or neurologic exams
* Speech discrimination < 60% in any ear

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change from the baseline in the Hearing In Noise Test (HINT) score at 6 months | at screening and 6 months after starting hearing aids use
  HINT measures a person's ability to hear speech in quiet and in noise. In the test, the patient is required to repeat sentences both in a quiet environment and with competing noise being presented from different directions.

SECONDARY OUTCOMES:
changes from the baseline in central auditory processing disorder test score at 1, 3, 6, 9 and 12 months | at screening, 1, 3, 6, 9, and 12 months after starting hearing aids use
  The central auditory processing disorder test is composed of three subtests; duration pattern test, frequency pattern test and dichotic words test. The patient is required to discriminate long duration sound from short one and high frequency sound from low one, and to repeat two words that are given simultaneously.
changes from the baseline in the HINT score at 3, 9, and 12 months | baseline, 3, 9 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jong Woo Chung, MD, Study Chair — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
Data is being analyzed.